CLINICAL TRIAL: NCT05486845
Title: The Effect of the Use of Lower Back Pillow.
Brief Title: Special Lower Back Pillow Examination
Acronym: LBP PILLOW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: SzegedU_LBP PILLOW
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain
Keywords: LBP; special pillow; lower back pillow
MeSH Terms: conditions — Low Back Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adults (Experimental): People who use the lower back pillow.
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — We are planning a questionnaire survey. We combine our own questions with validated, official questionnaires. Validated forms ask for an assessment of the extent of low back pain and the quality of experienced stress.

SUMMARY:
Low back pain is a significant, serious and widespread problem in our world today, both in terms of social and economic burdens. It should be emphasized that even the young adult age group is very often affected by non-specific, low back pain without proven pathoanatomical changes.

DETAILED DESCRIPTION:
We plan to examine the use of a special lower back pillow and the time period of the sitting position. We would like to know how it helps to prevent and treat low back pain. We would like to know more about the people's pillow usage habits.

We are planning a questionnaire survey. We combine our own questions with validated, official questionnaires. Validated forms ask for an assessment of the extent of low back pain and the quality of experienced stress.

ELIGIBILITY:
Inclusion Criteria:

* in case of patients with low back pain: chronic pain
* in case of asymptomatic individuals: no symptomes

Exclusion Criteria:

* serious neurologycal symptomes
* serious scoliosis
* previous surgery which affected the local stabilizers
* serious pulmonar disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
MEDICAL HISTORY RECORD SHEET | 3 minutes
  We created an individual patient examination form, in which we could ask our subjects about their lifestyle habits and about their low back pain.
THE QUEBEC BACK PAIN DISABILITY SCALE (QBPDS) | 2 minutes
  The Quebec back pain disability scale is a condition-specific questionnaire developed to measure the level of functional disability for patients with low back pain (LBP) is a condition-specific questionnaire developed to measure the level of functional disability for patients with low back pain (LBP). The original purpose of the questionnaire is to take into account the functional limitations related to pain, to monitor the progress of individual patients and to compare the evolution of LBP subjects incorporated in rehabilitation programs.
THE PERCEIVED STRESS SCALE (PSS) | 2 minutes
  The Perceived Stress Scale is a classic stress assessment instrument. The tool remains a popular choice for helping us understand how different situations affect our feelings and our perceived stress. The questions in this scale ask about your feelings and thoughts during the last month. In each case, you will be asked to indicate how often you felt or thought a certainn way.
VISUAL ANALOG SCALE | 1 minute
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. VAS is the most common pain scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Szeged, Csongrád-Csanád, Hungary

IPD SHARING:
Plan to Share IPD: Undecided